CLINICAL TRIAL: NCT00842894
Title: A Prospective, Multicentre, Open Label, Non-controlled, Observational, 26-week Study in Patients Using NovoMix® 30 (Biphasic Insulin Aspart 30) or Levemir® (Insulin Detemir) for Treatment of Type 2 Diabetes Mellitus in Macedonia
Brief Title: Safety of NovoMix® 30 or Levemir® for Treatment of Type 2 Diabetics in Macedonia
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3716
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Insulin detemir
  Interventions: Drug: insulin detemir
- Biphasic insulin aspart 30
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: insulin detemir — Safety and effectiveness data collection in connection with the use of the drug.
  Other Names: NN304; Levemir®
  Groups: Insulin detemir
Drug: biphasic insulin aspart 30 — Safety and effectiveness data collection in connection with the use of the drug in daily clinical practice.
  Groups: Biphasic insulin aspart 30

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to investigate the incidence of serious adverse drug reactions when using NovoMix® 30 (biphasic insulin aspart 30) or Levemir® (insulin detemir) for treatment of type 2 diabetes mellitus under normal clinical practice conditions in Macedonia.

ELIGIBILITY:
Inclusion Criteria:

* After the physician decision has been made to use biphasic insulin aspart 30 or insulin detemir therapy, any subject with Type 2 diabetes is eligible for the study, including newly-diagnosed subjects who have never received insulin or an insulin analogue before.Particular attention should be paid to the drug interactions that are listed within the product label

Exclusion Criteria:

* Subjects who are unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for the final visit
* Subjects currently being treated with biphasic insulin aspart 30 or insulin detemir
* Subjects who were previously enrolled in this study
* Subjects with a hypersensitivity to biphasic insulin aspart 30 or insulin detemir or to any of the excipients
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within next 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from speciality practice settings who have been deemed appropriate to receive biphasic insulin aspart 30 or insulin detemir as new treatment and as part of routine out-patient care by the prescribing physician.
Sampling Method: Non-Probability Sample
Enrollment: 3421 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse drug reactions (SADRs) | after 26 weeks

SECONDARY OUTCOMES:
Number of all minor hypoglycaemic events | during 4 weeks preceding each visit
Number of all major hypoglycaemic events | during 13 weeks preceding each visit
HbA1c | after 26 weeks
Percentage of subjects to reach HbA1c below 7.0% | after 13 weeks and 26 weeks
The effect on glycaemic control as measured by FPG (fasting plasma glucose) | after 13 weeks and 26 weeks
The effect on glycamic control as measured by PG profile | after 13 weeks and 26 weeks
Change in body weight | after 13 weeks and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Skopje, North Macedonia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com